CLINICAL TRIAL: NCT01526109
Title: Effect of Strength Training and Whole Body Vibration on Cognitive Function, Behavioral and Functional Capacity in Healthy Elderly.
Brief Title: Effect of Strength Training and Whole Body Vibration in Healthy Elderly
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was finished since the University has been closed
Sponsor: Universidade Gama Filho (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Andrea Camaz Deslandes, Principal investigator, Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 040.2011
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2012-02

CONDITIONS: Health Behavior
Keywords: elderly; quality of life; functional capacity; cognitive function; physical exercise
MeSH Terms: conditions — Health Behavior; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- strength training group (Experimental): Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of strength training twice a week consists of six exercises for major muscle groups: leg press, bench press, lat pull down, knee extension, knee flexion and Abdominal (3 sets of 10-12 repetitions at 60-80% of 1 RM with 3 min interval between sets and between workouts).
  Interventions: Behavioral: Strength training group
- Control group (Placebo Comparator): Participants will undergo a training program set for the three functional groups of ten minutes duration, followed by thirty minutes of functional exercises twice a week (2-3 sets of 30 sec. At intervals of 60 s between stimuli) carry out a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk without intensity
  Interventions: Behavioral: Control group
- whole-body vibration training group (Experimental): Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of exercise stimuli to whole-body vibration twice a week (2-3 sets of 30 sec. with frequency of stimulation at 30 Hz with 60 s intervals between stimuli), the platform will hold a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk.
  Interventions: Behavioral: Whole-body vibration training group

INTERVENTIONS:
Behavioral: Strength training group — Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of strength training twice a week consists of six exercises for major muscle groups: leg press, bench press, lat pull down, knee extension, knee flexion and Abdominal (3 sets of 10-12 repetitions at 60-80% of 1 RM with 3 min interval between sets and between workouts).
  Other Names: resistence training
  Arms: strength training group
Behavioral: Control group — Participants will undergo a training program set for the three functional groups of ten minutes duration, followed by thirty minutes of functional exercises twice a week (2-3 sets of 30 sec. At intervals of 60 s between stimuli) carry out a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk without intensity
  Other Names: no intensity
  Arms: Control group
Behavioral: Whole-body vibration training group — Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of exercise stimuli to whole-body vibration twice a week (2-3 sets of 30 sec. with frequency of stimulation at 30 Hz with 60 s intervals between stimuli), the platform will hold a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk.
  Other Names: WBV training
  Arms: whole-body vibration training group

SUMMARY:
Quality of Life (Qol) is a complex concept which relates to the perception of subjective satisfaction, especially in elderly population. It also relates to the self-perception of psychological status, independence level, to the social relationships, and to the environment where the elderly person lives. Consequently, there are a number of factors which may change the perception of QoL, namely the occurrence of diseases, physical impairment or incapacity, and the rupture of social relationship, as well as the aging process itself. Physical exercise is associated to improvement of mental and physical health. However, few studies investigated the effect of strength training and whole- body vibration training on elderly subjects. Following this line of reasoning, the purpose of the present study is to assess the effect of physical exercise on cognition and functional abilities in elderly subjects. Design: Randomized controlled trial, double-blinded, with 12-week follow-up. Setting: Gama Filho University. Participants: Healthy Elderly. Interventions: The patients will be randomly assigned to a strength training group (STG), whole-body vibration training group (WBVG) and a control group (CG). Main outcome measures: Cognitive function will be assessed using Mini Metal State Examination (MMSE), Trail A and B, Digit Span, Stroop Test, Rey auditory-verbal learning test and Clock Test, and functional capacity will be evaluated using Senior Fitness Test, American Alliance for Health, Physical Education, Recreation & Dance(AAHPERD)functional fitness test, and Short Form 36(SF-36) health survey.

DETAILED DESCRIPTION:
Design: Three-month controlled, randomized, and double-blind study. The subjects will be recruited from the Gama Filho University. They will be randomized with a blind design to a whole-body vibration training group (WBV), strength training group (STG) and control group (CG) by a researcher who will not participate of the initial assessments.

Intervention

The study is a longitudinal randomized clinical trial. The subjects will perform three visits to the laboratory where they will be submitted to neuropsychological, behavioral and physical evaluations. These evaluations will be performed before and after three months of training. Each visit will last about an hour and a half. After a period of one week of adaptation, subjects begin training with the charges set out in this study. All groups will carry out training twice a week, forty minutes, for three months. Next, will be described in detail the experimental procedures in each group:

STG Group Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of strength training twice a week consists of six exercises for major muscle groups: leg press, bench press, lat pull down, knee extension, knee flexion and Abdominal (3 sets of 10-12 repetitions at 60-80% of 1 RM with 3 min interval between sets and between workouts).

WBV Group Participants will undergo a training program set for the three functional groups, which lasted ten minutes, followed by thirty minutes of exercise stimuli to whole-body vibration training twice a week (2-3 sets of 30 sec. with frequency of stimulation at 30 Hz with 60 s intervals between stimuli), the platform will hold a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk.

Control Group Participants will undergo a training program set for the three functional groups of ten minutes duration, followed by thirty minutes of functional exercises twice a week (2-3 sets of 30 sec. At intervals of 60 s between stimuli) carry out a range of six functional exercises combining squats and isometric or dynamic exercises for the upper limbs and trunk without intensity.

ELIGIBILITY:
Inclusion Criteria:

* elderly (> 60 years)
* without diagnosis of mental illness or cognitive decline
* literate
* have not committed to physical exercises.

Exclusion Criteria:

* scored outside the cutoff point set in the scales of depressive symptoms (Beck > 18)
* cognitive decline (MSSE < 18 for low educational level and < 24 for high school).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Short Form 36 (SF-36) questionaire at 12 weeks | from date to randomization at 12 weeks
  The quality of life questionnaire Short Form 36 (SF-36) is multidimensional, consisting of 36 items, divided into eight scales, each scale assesses a health concept, they are: limitations in physical activities because of health problems, limitations in social activities due to physical or emotional problems, limitations in daily activities due to health problems, body pain, mental health, limitations in daily activities due to emotional problems, vitality (energy and fatigue), perception of general health.

SECONDARY OUTCOMES:
Change from baseline in Senior Fitness Test at 12 weeks | from date to randomization at 12 weeks
  The assessment of functional capacity of patients will be conducted through the battery functional tests of the Senior Fitness Test. Will be evaluated regarding their balance, strength, lower limb and upper, flexibility, agility, running and cardiovascular fitness. The battery consists of seven physical tests: 1) Time to Up and Go (TUG), 2) get up and down, 3) flexibility and 4) strength of MI and MS, 5) 6-minute walk, 6) sit down and test achieve, and 7) test bench.
Change from baseline in American Alliance for Health, Physical Education, Recreation & Dance(AAHPERD)functional fitness test at 12 weeks | from date to randomization at 12 weeks
  The participant begins the test in a chair with your heels flat on the floor. At the signal of "ready now" moves to the right and around a cone positioned at 1.50 m and 1.80 m behind to the side of the chair, returning to his chair and sat down. Immediately the participant gets up, moves to the left and around the second cone, returning to his chair and sat down again. So complete a circuit. The individual must complete two full circuits.
Change from baseline in Trail Making Test at 12 weeks | from date to randomization at 12 weeks
  Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters. The patient should be instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper.
Change from baseline in Mini Metal State Examination (MMSE) at 12 weeks | from date to randomization at 12 weeks
  The MMSE is a brief screening test for cognitive capabilities that evaluates orientation (spatial and time), attention, concentration, memory, calculation, language, and praxis. The score ranges from 0 to 30, with higher scores indicating better performance.
Change from baseline in Digit Test at 12 weeks | from date to randomization at 12 weeks
  A series of number sequences are presented to the subject. In the first portion of the test, the subject is asked to reproduce the exact sequence, whereas in the second portion he/she is asked to repeat the sequence backwards. The Digit span evaluated attention, concentration and working memory.
change from baseline in Stroop Test at 12 weeks | from date to randomization at 12 weeks
  There are three parts to the test. In Part 1, the subject must name the colors painted (blue, green, red and yellow) in a card. In Part 2, the subject reads the color names (blue, green, red and yellow) painted ignoring the printed words. In Part 3, the subject must name the color (blue, green, red and yellow) painted, ignoring the color name printed on the card, which is always different color painted.
Change from baseline in Rey Complex Figure Test at 16 weeks | from date to randomization at 12 weeks
  It uses a complex geometric figure. The examinee is asked to copy the figure with as many details in a white paper in a horizontal position.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Deslandes, Dr, Principal Investigator — UGF
Locations (1):
- Universidade Gama Filho, Rio de Janeiro, Rio de Janeiro, Brazil